CLINICAL TRIAL: NCT05291845
Title: Candida Antigen and Bivalent HPV Vaccine in the Treatment of Multiple Warts: Monotherapy Versus Combined Therapy
Brief Title: Candida Antigen and Bivalent HPV Vaccine in the Treatment of Multiple Warts
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Essam, Lecturer of Dermatology, Zagazig University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: C.ag-vs-B.HPV.V
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-04

CONDITIONS: Warts; Human Papilloma Virus
MeSH Terms: conditions — Warts | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Candida antigen group (Experimental): 54 patients will be treated with Candida antigen. All patients will be directly injected with Candida antigen into the largest wart using an insulin syringe. Injections will be done at 2-week intervals until complete clearance will be achieved or for a maximum of five treatment sessions.
  Interventions: Biological: Candida antigen vaccine
- Bivalent HPV vaccine (Experimental): 54 patients will be treated with the Bivalent HPV vaccine. All patients will be directly injected with the vaccine into the largest wart using an insulin syringe. Injections will be done at 2-week intervals until complete clearance will be achieved or for a maximum of five treatment sessions.
  Interventions: Biological: Bivalent HPV vaccine
- both agents group (Experimental): 54 patients will be treated with Both agents at the same session. Injections will be done at 2-week intervals until complete clearance will be achieved or for a maximum of five treatment sessions.
  Interventions: Biological: Candida antigen vaccine; Biological: Bivalent HPV vaccine

INTERVENTIONS:
Biological: Candida antigen vaccine — we will study the efficacy and safety of agent in the treatment of multiple warts, we will follow up the recurrence rate of each group
  Arms: Candida antigen group; both agents group
Biological: Bivalent HPV vaccine — we will study the efficacy and safety of agent in the treatment of multiple warts, we will follow up the recurrence rate of each group
  Arms: Bivalent HPV vaccine; both agents group

SUMMARY:
To follow up the efficacy and safety of Candida antigen, bivalent HPV vaccine in treatment of common warts either mono or combined intralesional therapy

DETAILED DESCRIPTION:
* Group A: 54 patients will be treated with Candida antigen. All patients will be directly injected with Candida antigen into the largest wart using an insulin syringe. Injections will be done at 2-week intervals until complete clearance will be achieved or for a maximum of five treatment sessions.
* Group B: 54 patients will be treated with bivalent HPV vaccine solution intralesional into the largest wart using an insulin syringe. Injections will be done at 2-week intervals until complete clearance will be achieved or for a maximum of five treatment sessions.
* Group C: 54 patients will be treated with both agents intralesionally into the largest wart using an insulin syringe at 2-week intervals until complete clearance will be achieved or for a maximum of five treatment sessions.

it is thought that candida antigen act through a cell-mediated immune response and bivalent HPV vaccine act mainly through humoral immunity, so we want to study their effect as single or mixed agents

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple, recalcitrant, or non-recalcitrant common warts of different sites, sizes, duration, and with or without distant lesions will be enrolled in the study

Exclusion Criteria:

* Pregnant female. Hypersensitivity to Candida antigen or bivalent HPV vaccine

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2022-04-03 (Actual); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
complete response | upto 3 months
  if there is disappearance of warts and return of the normal skin markings
partial response | upto 3 months
  if warts regressed in size by 50-99% (the size will be measured as the summation of size of all lesions in cm)
no response | upto 3 months
  if there is < 50% decrease in wart size. (the size will be measured as the summation of size of all lesions in cm)

SECONDARY OUTCOMES:
recurrence rate after recovery | follow up for 6 months after recovery
  appearance of new lesions or recurrence of previous one

CONTACTS AND LOCATIONS:
Overall Officials: Reham Essam, MD, Principal Investigator — Zagazig University; Ahmad Nofal, MD, Study Director — Zagazig University
Locations (1):
- Reham Essam, Zagazig, Al Sharqia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nofal A, Marei A, Ibrahim AM, Nofal E, Nabil M. Intralesional versus intramuscular bivalent human papillomavirus vaccine in the treatment of recalcitrant common warts. J Am Acad Dermatol. 2020 Jan;82(1):94-100. doi: 10.1016/j.jaad.2019.07.070. Epub 2019 Jul 29. PMID 31369771
- [Background] Nassar A, Alakad R, Essam R, Bakr NM, Nofal A. Comparative efficacy of intralesional Candida antigen, intralesional bivalent human papilloma virus vaccine, and cryotherapy in the treatment of common warts. J Am Acad Dermatol. 2022 Aug;87(2):419-421. doi: 10.1016/j.jaad.2021.08.040. Epub 2021 Aug 28. No abstract available. PMID 34464624
- See also: Intralesional versus intramuscular bivalent human papillomavirus vaccine in the treatment of recalcitrant common warts — https://doi.org/10.1016/j.jaad.2019.07.070
- See also: Comparative efficacy of intralesional Candida antigen, intralesional bivalent human papilloma virus vaccine, and cryotherapy in the treatment of common warts — https://doi.org/10.1016/j.jaad.2021.08.040